CLINICAL TRIAL: NCT03410537
Title: A Randomized, Double-blind, Placebo Controlled Clinical Trial Comparing Effects of Taurine Supplementation on Lower Extremity Vasculopathy in Patients With Diabetes
Brief Title: Taurine Supplementation on Lower Extremity Vasculopathy in Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, MD,PhD,Director, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSLEVD
Record Dates: First submitted 2017-12-28; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Taurine; Diabetes; Lower Extremity Artery Disease
MeSH Terms: conditions — Diabetes Mellitus | interventions — Taurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Taurine Supplementation (Experimental): Taurine 2.4mg/d for 12 weeks
  Interventions: Drug: Taurine
- Placebo (Placebo Comparator): Placebo 2.4mg/d for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Taurine
  Arms: Taurine Supplementation
Drug: Placebo
  Arms: Placebo

SUMMARY:
Diabetes has become important risk factors for threatening human life and health. Lower extremity arterial occlusive are the common complications of diabetes.Sulfur amino acid is the indispensable amino acid in mammals, and its metabolites include Taurine, Hydrogen sulfide (H2S) and sulfur dioxide (SO2). Taurine was first isolated more than 150 years ago from ox (Taurus) bile. Although the taurine can be synthesized in vivo by cysteine in the presence of cysteine dioxygenase, it is mainly acquired from dietary sources, such as eggs, meat, and seafood. H2S is a biologically relevant mediator and plays potential roles in several physiological processes and disease states in the body. H2S is synthesized from 2 sulfur-containing amino acids, l-cysteine andl-methionine, by the 3 enzymes,cystathionine-γ-lyase (CSE), cystathionine-β-synthetase(CBS), and3-mercaptopyruvate sulfurtransferase (3-MST). Previous studies have demonstrated that Taurine and H2S may play important roles in the development of the microangiopathy and lower extremity arterial occlusive.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age between 18-80 years old
2. Type 2 diabetes

Exclusion Criteria:

1. Type2 diabetes with acute diabetic complications.
2. Type1 diabetes.
3. History of cardio-cerebral vascular events, such as congestive heart failure, myocardial infarction or stroke within 3 months.
4. Hypohepatia (AST or AST is twice higher than the upper limit) or history of hepatitis or cirrhosis, hepatic encephalopathy.
5. Renal insufficiency (serum creatinine 1.5 times higher than the upper limit) or history of dialysis and nephritic syndrome.
6. Acute infections, tumor, severe arrhythmia, mental disorders, alcohol or medicine addiction.
7. Fertile woman without contraceptives.
8. Any surgical or medical conditions that significantly influence absorption, distribution, metabolism or excretion of the intervention drugs.
9. Allergic to or have contraindication to the intervention drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Ankle-brachial index | Baseline, 12weeks(End of Trial)
  Changes of ankle-brachial index after 12 weeks.

SECONDARY OUTCOMES:
24-hours mean blood pressure. | Baseline, 12weeks(End of Trial)
Pulse wave velocity(PWV) | Baseline, 12weeks(End of Trial)
Fasting plasma glucose | Baseline, 12weeks(End of Trial)
HbA1c | Baseline, 12weeks(End of Trial)
Lipid profile (triglyceride, total cholesterol, LDL-c; HDL-c; mmol/L) | Baseline, 12weeks(End of Trial)
Carotid intima-media thickness(IMT) | Baseline, 12weeks(End of Trial)
Body mass index(BMI) | Baseline, 12weeks(End of Trial)
Fasting serum insulin | Baseline, 12weeks(End of Trial)

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No